CLINICAL TRIAL: NCT01014286
Title: Lung Cancer Mutation Consortium Protocol
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-0756.cc; RC2CA148394 (NIH)
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Adenocarcinoma of Lung, Stage IV
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsy remnant tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced Adenocarcinoma: Stage IV adenocarcinoma who have undergone biopsy with remnant tissue.

SUMMARY:
The primary objective of this protocol is to determine the frequency of oncogenic mutations in 1000 patients with advanced adenocarcinoma of the lung. The linked clinical and mutational analyses will be used to determine the frequency of each mutation, its association with clinical features and outcome, and its association with other mutations. As future therapeutic protocols specific for these mutations are developed, patients may be notified of their eligibility for these studies. Future translational studies may be used to: a) unravel the complex biology of lung cancer; b) identify prognostic markers; c) define predictive markers of response/resistance to new therapies; d) identify new targets. A secondary goal is to establish a consortium of sites that have the capability of conducting multiple mutation testing in a Clinical Laboratory Improvement Amendments (CLIA) certified lab.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (=> 18 years of age) who are undergoing further evaluation for the diagnosis or treatment of advanced adenocarcinoma of the lung.
2. Diagnosed May 2012 or later
3. Oral and written informed consent.

Exclusion Criteria:

1. Lung cancer histologies other than adenocarcinoma
2. Lack of adequate tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV adenocarcinoma of the lung who have undergone biopsy with remnant tissue
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2009-09-16; Primary Completion 2016-09-01 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
Frequency of oncogenic mutations in patients with advanced adenocarcinoma of the lung. | Five years
  The primary objective of this protocol is to determine the frequency of oncogenic mutations in patients with advanced adenocarcinoma of the lung.
Rate of oncogenic mutations in patients with advanced adenocarcinoma of the lung. | Five years
  The primary endpoint of this protocol is the mutation rate.

SECONDARY OUTCOMES:
Associations between each mutation and clinical outcomes. | Two years
  The secondary objectives of this protocol are to study the associations between each mutation and clinical outcomes, e.g., survival, clinical features, e.g. smoking status, age, and other mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bunn, M.D., Study Director — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kris MG, Johnson BE, Berry LD, Kwiatkowski DJ, Iafrate AJ, Wistuba II, Varella-Garcia M, Franklin WA, Aronson SL, Su PF, Shyr Y, Camidge DR, Sequist LV, Glisson BS, Khuri FR, Garon EB, Pao W, Rudin C, Schiller J, Haura EB, Socinski M, Shirai K, Chen H, Giaccone G, Ladanyi M, Kugler K, Minna JD, Bunn PA. Using multiplexed assays of oncogenic drivers in lung cancers to select targeted drugs. JAMA. 2014 May 21;311(19):1998-2006. doi: 10.1001/jama.2014.3741. PMID 24846037